CLINICAL TRIAL: NCT01607515
Title: Non Invasive Measurement of Cardiac Index by Impedance Cardiography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Graz (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 24-205 ex 11/12
Record Dates: First submitted 2012-04-13; First posted 2012-05-30 (Estimated); Last update posted 2015-09-09 (Estimated); Status verified 2015-09

CONDITIONS: Pulmonary Hypertension
Keywords: Pulmonary hypertension; Cardiac index; impedance cardiography
MeSH Terms: conditions — Hypertension, Pulmonary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- suspected PH (Other): Patients who undergo right heart catheterization for PH diagnosis undergo impedance cardiography
  Interventions: Other: Impedance cardiography

INTERVENTIONS:
Other: Impedance cardiography — noninvasive measure of cardiac index by impedance cardiography.
  Other Names: patients with a clinical suspicion of PH

SUMMARY:
Pulmonary hypertension (PH) is defined as a pulmonary arterial mean pressure (meanPAP) ≥ 25 mmHg in the right heart catheterization.

There are different forms of PH defined in the classification of Dana Point 2008.

PH is diagnosed with right heart catheterization but there are other non invasive methods which can be used for screening like echocardiography, stress echocardiography and cardio pulmonary exercise testing.

For prognosis of PH patients the limitation of the pulmonary circulation is very important. Therefore the cardiac index (CI) is a good parameter for the right ventricular function. The gold standard for CI measures is the thermodilution, an invasive method performed during right heart catheterization.

DETAILED DESCRIPTION:
In this study the investigators want to evaluate the impedance cardiography (ICG) as a non invasive method for CI measurement. An alternating current of max 400µA and 45 kHz is conducted through the body. The way of the smallest resistance is the blood in the aorta. The impedance changes with the pulsatile blood flow. Out of the Impedance change there can be calculated the CI.

ELIGIBILITY:
Inclusion Criteria:

* patients who have right heart catheterization written informed consent

Exclusion Criteria:

* patients who don't have right heart catheterization no written informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Comparison of CI measured by ICG and Thermodilution | recruitment over 1.5 year (Data collection), followed by data analysis and interpretation (overall 2 yearsfrom start of recruitment)
  assessment of the Specificity and sensitivity of ICG for CI measurement

CONTACTS AND LOCATIONS:
Overall Officials: Horst Olschewski, MD, Principal Investigator — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria